CLINICAL TRIAL: NCT07048561
Title: Changes in Health-related Physical Fitness on the Behavioural and Electrophysiological Aspects of Cool and Hot Executive Function in Older Adults: A Prospective Study
Brief Title: Health-related Physical Fitness and Executive Function in Older Adults: A Prospective Study
Status: Recruiting | Type: Observational
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Principal Investigator, Ruei-Hong Li, Doctoral student, National Taiwan Normal University
Other Study IDs: NTNU_PACNL_HPF_EF_P
Record Dates: First submitted 2025-05-21; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Older Adults (65 Years and Older); Fitness Testing; Executive Function (Cognition); Prospective Study; Event-Related Potentials
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older adults: Older adults aged 65 and above.
  Interventions: Other: observation alone

INTERVENTIONS:
Other: observation alone — No interventions will be conducted during the one-year observation period, maintaining participants' normal daily living conditions.
  Other Names: one-year observation

SUMMARY:
This study aims to explore the relationship between health-related physical fitness and behavioural and electrophysiological aspects of cool and hot executive function in older adults through a year prospective study design. The main questions it aims to answer whether changes in health-related physical fitness will positively predict changes in behavioural and electrophysiological aspects of cool and hot executive functions in older adults. The participants will be asked to complete pre-test, a one-year observation period, and post-test. Both pre- and post-tests will measure health-related physical fitness, executive function, and various demographic variables and covariates. Health-related physical fitness assessments include cardiorespiratory endurance (YMCA submaximal cycle test), muscular strength (grip strength, chest press, and leg press), muscular endurance (30-second chair stand, 30-second bicep curl), flexibility (range of motion), and balance (Balance Error Scoring System). Executive function will be measured using the Stroop test and emotional Stroop test, with concurrent EEG recording of brain activity. Demographic variables and covariates include sex, age, years of education, annual income, Pittsburgh Sleep Quality Index (PSQI), International Physical Activity Questionnaire (IPAQ) Taiwan short form, World Health Organisation Quality of Life Brief Assessment (WHOQOL-BREF) Taiwan version, Geriatric Depression Scale, Mini-Mental State Examination (MMSE), digit span tests, and step count recorded by mobile phones or watches over the previous month, resting heart rate, and resting blood pressure. No interventions will be conducted during the one-year observation period, maintaining participants' normal daily living conditions.

DETAILED DESCRIPTION:
Executive function refers to higher-order cognitive functions responsible for planning, organisation, and problem-solving. These functions decline with age and are crucial for maintaining independence and quality of life in older adults. Research indicates that health-related physical fitness may serve as a protective factor against executive function decline, encompassing cardiorespiratory endurance, body composition, muscular strength, muscular endurance, flexibility, and balance. However, no studies have simultaneously tracked the relationship between these health-related physical fitness components and executive function. Thus, this study employs a one-year prospective design to investigate the relationship between changes in health-related physical fitness and executive function in older adults. The study will recruit 200 older adults aged 65 or above for pre-test, a one-year observation period, and post-test. Both pre- and post-tests will measure health-related physical fitness, executive function, and various demographic variables and covariates. Health-related physical fitness assessments include cardiorespiratory endurance (YMCA submaximal cycle test), muscular strength (grip strength, chest press, and leg press), muscular endurance (30-second chair stand, 30-second bicep curl), flexibility (range of motion), and balance (Balance Error Scoring System). Executive function will be measured using the Stroop test and emotional Stroop test, with concurrent EEG recording of brain activity. Demographic variables and covariates include sex, age, years of education, annual income, Pittsburgh Sleep Quality Index (PSQI), International Physical Activity Questionnaire (IPAQ) Taiwan short form, World Health Organisation Quality of Life Brief Assessment (WHOQOL-BREF) Taiwan version, Geriatric Depression Scale, Mini-Mental State Examination (MMSE), digit span tests, and step count recorded by mobile phones or watches over the previous month, resting heart rate, and resting blood pressure. No interventions will be conducted during the one-year observation period, maintaining participants' normal daily living conditions. This study will provide preliminary evidence on the relationship between health-related fitness and executive function, offering guidance to the public and government agencies for developing exercise programmes aimed at enhancing executive function. By understanding key health-related physical fitness components for exercise design, Taiwan, which faces an ageing society, may potentially reduce government financial and social burdens related to dementia care.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or above.
* Able to engage in fitness testing.
* Normal vision or corrected-to-normal vision.

Exclusion Criteria:

* Suffering from cardiopulmonary-related diseases.
* Suffering from cognitive, neurological or psychiatric disorders (e.g., dementia, Parkinson's disease, epilepsy, depression, schizophrenia, etc.).
* Suffering from infectious diseases (e.g., hepatitis, human immunodeficiency virus or Creutzfeldt-Jakob disease).
* Having a history of drug or alcohol abuse.
* Having colour vision deficiency (e.g., colour blindness).
* Having a family history of aneurysm.
* Taking medications that affect brain function.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Study population are older adults aged 65 or above.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Health-related physical fitness (cardiorespiratory endurance) | From enrolment to the end of observation at one year.
  Cardiorespiratory endurance was assessed using the YMCA Submaximal Cycle Ergometer Test. The protocol comprised four 3-minute stages at 50 rpm, beginning with a 25W workload in stage one. Stage two workload was determined by steady-state heart rate (HR) achieved during the final two minutes of stage one (tolerance ±5 beats/min): <80 beats/min = 125W; 80-89 beats/min = 100W; 90-100 beats/min = 75W; >100 beats/min = 50W. Stages three and four increased workload by 25W increments, targeting two consecutive steady-state HRs between 110 beats/min and 85% HRmax. Stage duration was extended by one-minute intervals when steady-state criteria were not met (HR variation >5 beats/min or <110 beats/min during final two minutes). Peak VO₂ was estimated using established formulae.
Health-related physical fitness (muscular strength) | From enrolment to the end of observation at one year.
  Muscular strength was assessed by handgrip strength, chest press, and leg press. Hand grip strength was assessed using a digital hand dynamometer. Chest and leg press was assessed using chest and leg press machines, respectively, following a standardised four-stage protocol. Participants initially performed 10-12 repetitions at minimal resistance for familiarisation and warm-up. Subsequently, they completed 5-10 repetitions with progressively increasing resistance (5-10% increments for upper body; 10-20% for lower body), with 3-5 minute rest intervals between attempts. This process continued until participants could perform fewer than five repetitions. The final successfully completed workload served as the basis for one-repetition maximum (1-RM) estimation using established conversion tables.
Health-related physical fitness (muscular endurance) | From enrolment to the end of observation at one year.
  Muscular endurance was assessed using the 30-second bicep curl and 30-second chair stand from the Senior Fitness Test. The 30-second bicep curl required participants to sit upright on the chair edge, favouring their dominant side, with feet flat on the ground. Using a handshake grip, they held a dumbbell (5 pounds for females, 8 pounds for males) in their dominant hand, with the arm initially hanging straight down beside the chair. Complete arm flexion and extension constituted one repetition, with participants instructed to perform maximal repetitions within 30 seconds. The 30-second chair stand required participants to sit centrally with backs straight, feet flat on the ground, and arms crossed over their chests. They performed maximal repetitions of standing up and sitting down within 30 seconds. The total number of repetitions in each test served as the respective muscular endurance indicator.
Health-related physical fitness (flexibility) | From enrolment to the end of observation at one year.
  Flexibility was assessed using range of motion measurements obtained with a joint goniometer. The goniometer's fulcrum was positioned at the centre of the target joint, with arms aligned to the bony landmarks of the proximal and distal segments. The resulting angular measurement represented the joint's range of motion.
Health-related physical fitness (balance) | From enrolment to the end of observation at one year.
  Balance was assessed using the Balance Error Scoring System (BESS). Participants maintained six stances for 20 seconds each with eyes closed and hands on hips: double-leg stance, single-leg stance on the non-dominant foot, and tandem stance with the non-dominant heel against the dominant toe. These three positions were performed on both a firm surface and a medium-density foam pad (45 cm × 45 cm × 13 cm).
  Errors were recorded for removing hands from hips, opening eyes, stepping, excessive hip movement (>30°), or lifting the foot. Each trial was scored with a maximum of 10 errors, with participants unable to maintain stance for 5 seconds receiving the maximum score. The total BESS score represented cumulative errors across all six conditions.
Executive function | From enrolment to the end of observation at one year.
  Executive function will be measured using the Stroop test and emotional Stroop test, with concurrent EEG recording of brain activity.

SECONDARY OUTCOMES:
Demographic questionnaire | From enrolment to the end of observation at one year.
  Demographic questionnaire include sex, age, years of education, and step count recorded by mobile phones or watches over the previous month.
Sleep quality (Pittsburgh Sleep Quality Index, PSQI) | From enrolment to the end of observation at one year.
  Sleep quality was assessed using the Pittsburgh Sleep Quality Index (PSQI), a validated self-report questionnaire comprising 19 items that evaluate sleep patterns over the preceding month. The instrument generates seven component scores: subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, sleep medication use, and daytime dysfunction. Each component is scored from 0 to 3, yielding a global score ranging from 0 to 21. Scores ≤5 indicate good sleep quality, whilst scores >5 suggest poor sleep quality, with higher values reflecting greater sleep impairment.
Physical activity (Taiwan version of the International Physical Activity Questionnaire, IPAQ) | From enrolment to the end of observation at one year.
  Physical activity was assessed using the Taiwan version of the International Physical Activity Questionnaire (IPAQ). This seven-item instrument measures metabolic equivalents (METs) across work, household, leisure, and sedentary activities over a seven-day period, expressed in kcal/kg/min. Activities are categorised as vigorous, moderate, and light intensity (walking), alongside sedentary behaviour, with frequency (days/week) and duration (minutes/session) recorded for each intensity level.
Quality of life (Taiwan version of World Health Organisation Quality of Life Brief Assessment, WHOQOL-BREF) | From enrolment to the end of observation at one year.
  Quality of life was assessed using the Taiwan version of the World Health Organization Quality of Life Questionnaire-Brief Form (WHOQOL-BREF), a validated 24-item instrument utilising a five-point Likert scale. Participants evaluated their experiences and perceptions over the preceding two weeks across four domains: physical health, psychological health, social relationships, and environmental factors. Two additional items assessed overall quality of life and general health satisfaction. This instrument provides comprehensive multidimensional assessment suitable for clinical and research applications.
Depressive symptoms (Geriatric Depression Scale) | From enrolment to the end of observation at one year.
  The Geriatric Depression Scale (GDS-15) comprises 15 items designed to assess depressive symptoms in older adults. Scores range from 0-15, with higher values indicating greater depressive symptomatology. Clinical cut-off points are established as follows: scores of 0-4 indicate normal mood, 5-8 suggest mild depression, 9-11 indicate moderate depression, and scores ≥12 suggest severe depression.
Cognitive function (Mini-Mental State Examination, MMSE) | From enrolment to the end of observation at one year.
  The Mini-Mental State Examination (MMSE) is a widely utilised cognitive screening instrument that provides quantitative assessment of cognitive function. This 30-item assessment evaluates multiple cognitive domains: orientation (10 points), memory encoding (3 points), attention and calculation (5 points), recall (3 points), and language with visuospatial construction (9 points). Total scores range from 0 to 30, with scores below 25 indicating potential cognitive impairment.
Working memory (Digit Span Tests) | From enrolment to the end of observation at one year.
  Working memory was assessed using the Digit Span subtest from the Wechsler Adult Intelligence Scale-Third Edition (WAIS-III). The subtest comprises forward digit sequences (16 items) and backward digit sequences (14 items), administered orally without written aids. Participants were required to reproduce number sequences verbally, either in the original order (forward condition) or in reverse order (backward condition). Each correct response received one point, yielding maximum possible scores of 16 and 14 points for the forward and backward conditions, respectively.
Resting heart rate | From enrolment to the end of observation at one year.
  Resting heart rate was measured using the Polar H10 chest-worn heart rate monitor. Participants were seated in a quiet, temperature-controlled environment for a minimum of five minutes prior to measurement to ensure cardiovascular stabilisation. Heart rate data were recorded continuously over a three-minute period.
Resting blood pressure | From enrolment to the end of observation at one year.
  Resting blood pressure was assessed using an automated oscillometric sphygmomanometer. Measurements were taken from the participant's non-dominant arm following a standardised protocol, with participants seated upright and feet flat on the floor.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Kai Chang, PhD, Study Director — National Taiwan Normal University; Ruei-Hong Li, MS, Principal Investigator — National Taiwan Normal University
Locations (1):
- National Taiwan Normal University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided